CLINICAL TRIAL: NCT01660321
Title: A Single Treatment, Pharmacokinetic (PK) and Tolerance Study of Natroba (Spinosad) Topical Suspension, 0.9% in Pediatric Subjects 6 Months to 4 Years of Age With an Active Head Lice Infestation
Brief Title: Pharmacokinetic (PK) and Tolerance Study of Natroba Topical Suspension in Pediatrics With an Active Head Lice Infestation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ParaPRO LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SPN-109-11
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Pediculosis
Keywords: Pediculosis capitis; Head Lice
MeSH Terms: conditions — Lice Infestations | interventions — spinosad; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Natroba (Experimental): Natroba (Spinosad) Topical Suspension, 0.9%
  Interventions: Drug: spinosad

INTERVENTIONS:
Drug: spinosad — A sufficient amount of Natroba Topical Suspension was applied to completely cover the scalp, worked out to the ends of the hair, and left in place for 10 minutes (±30 seconds), followed by a complete rinse and shampoo.
  Other Names: Natroba (spinosad) Topical Suspension, 0.9%

SUMMARY:
A pharmacokinetic and tolerance study of Natroba (spinosad) Topical Suspension, 0.9% in pediatric subjects 6 months to 4 years of age with an active head lice infestation.

DETAILED DESCRIPTION:
A Postmarketing Requirement Protocol, multicenter, open-label study in pediatric subjects 6 months to 4 years of age with an active head lice infestation designed to determine the topical absorption and safety of Natroba (spinosad) Topical Suspension, 0.9% for a single, 10 minute treatment for spinosad (Spinosyn A and Spinosyn D) and benzyl alcohol.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 6 months to 4 years of age.
2. Subjects must have had an active lice infestation including live lice.
3. Individuals in otherwise good general health, free of any systemic or dermatologic disorders which, in the opinion of the Principal Investigator or designee, would interfere with the study results or increase the risk of adverse events.
4. A parent (or guardian) must have signed an Informed Consent Form to allow any child to participate in the study.
5. Subjects must have been available to stay in the clinic for blood draws. Parents or guardians must have been available to stay in the clinic, with the subject, for the entire duration of the study.
6. Subjects must have had veins capable of insertion of a Heplock catheter or withstanding multiple blood draws as determined by the Principal Investigator or qualified phlebotomist.
7. Normal values (at screening) for serum chemistry and hematology for subjects, unless the principal Investigator or qualified medical designee determined that the abnormal value was not clinically significant.

Exclusion Criteria:

1. History of irritation or sensitivity to pediculicide or hair care products or ingredients.
2. History of known allergy or sensitivity to topical anesthetics including lidocaine and prilocaine.
3. History of allergy or sensitivity to Heparin.
4. Systemic diseases that could have interfered with the results of this study as determined by the Principal Investigator or designee.
5. Any condition or illness that, in the opinion of the Investigator or designee, may have compromised the objective of the protocol or the safety of the subject.
6. The use of antibiotics or other systemic medications within 2 weeks of the screening visit, which in the opinion of the Investigator or designee could have interfered with the outcome of the study.
7. Participation in a previous drug study within the past 30 days.
8. Individuals with any visible skin/scalp condition (other than from an active lice infestation) at the treatment site which would have interfered with the evaluations according to the opinion of the Investigator or designee.
9. Parents or guardians who, in the opinion of the Investigator, did not understand their child's requirements for study participation and/or may be likely to exhibit poor compliance.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dowling B Stough, M.D., Principal Investigator — Burke Pharmaceutical Research; Jeffrey C Seiler, M.D., Principal Investigator — Lice Solutions Resource Network, Inc.
Locations (2):
- United States (2):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Lice Solutions Resource Network, Inc., West Palm Beach, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall Study
Period: Overall Study
Arm/Group | Natroba
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Natroba
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 2 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Cmax for Spinosyn A
Description: Peak Plasma Concentration of Spinosyn A in Natroba (spinosad) Topical Suspension, 0.9%
Time Frame: Blood samples collected up to 12 hours post treatment - 0 (pre-treatment), 0.5, 1.0, 3.0, 6.0 and 12 hours post-treatment.
Population: Per Protocol. For all but 1 subject (Subject 02-202), all spinosyn A and spinosyn D concentrations were Below Quantification Level (BQL) or < 3.0 ng/mL for all samples. Therefore, Cmax, Tmax, and AUC 0-12 were not summarized.
Measure: Number; unit: ng/mL
Arm/Group | Natroba
Number analyzed (Participants) | 26
ng/mL | NA — For all but 1 subject (Subject 02-202), all spinosyn A and spinosyn D concentrations were Below Quantification Level (BQL) or < 3.0 ng/mL for all samples.

2. Primary Outcome: Tmax for Spinosyn A
Description: The time after administration of Natroba (spinosad) Topical Suspension, 0.9% when the maximum plasma concentration is reached for Spinosyn A.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: hours
Arm/Group | Natroba
Number analyzed (Participants) | 26
hours | NA — For all but 1 subject (Subject 02-202), all spinosyn A and spinosyn D concentrations were Below Quantification Level (BQL) or < 3.0 ng/mL for all samples.

3. Primary Outcome: AUC (0-12) for Spinosyn A
Description: Area under the plasma concentration versus time curve (AUC) of Spinosyn A in Natroba (spinosad) Topical Suspension, 0.9%.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: ng*hr/mL
Arm/Group | Natroba
Number analyzed (Participants) | 26
ng*hr/mL | NA — For all but 1 subject (Subject 02-202), all spinosyn A and spinosyn D concentrations were Below Quantification Level (BQL) or < 3.0 ng/mL for all samples.

4. Primary Outcome: Cmax for Spinosyn D
Description: Peak Plasma Concentration of Spinosyn D in Natroba (spinosad) Topical Suspension, 0.9%
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: ng/mL
Arm/Group | Natroba
Number analyzed (Participants) | 26
ng/mL | NA — For all but 1 subject (Subject 02-202), all spinosyn A and spinosyn D concentrations were Below Quantification Level (BQL) or < 3.0 ng/mL for all samples.

5. Primary Outcome: Tmax for Spinosyn D
Description: The time after administration of Natroba (spinosad) Topical Suspension, 0.9% when the maximum plasma concentration is reached for Spinosyn D.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: hours
Arm/Group | Natroba
Number analyzed (Participants) | 26
hours | NA — For all but 1 subject (Subject 02-202), all spinosyn A and spinosyn D concentrations were Below Quantification Level (BQL) or < 3.0 ng/mL for all samples.

6. Primary Outcome: AUC (0-12) for Spinosyn D
Description: Area under the plasma concentration versus time curve (AUC) of Spinosyn D in Natroba (spinosad) Topical Suspension, 0.9%.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: ng* hr/mL
Arm/Group | Natroba
Number analyzed (Participants) | 26
ng* hr/mL | NA — For all but 1 subject (Subject 02-202), all spinosyn A and spinosyn D concentrations were Below Quantification Level (BQL) or < 3.0 ng/mL for all samples.

7. Primary Outcome: Cmax for Benzyl Alcohol
Description: Peak Plasma Concentration of benzyl alcohol (above Limit of Quantitation (1.0 μg/mL) in Natroba (spinosad) Topical Suspension, 0.9%.
Time Frame: as for outcome 1
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Natroba
Number analyzed (Participants) | 26
μg/mL | 1.123 (0.3071) [0.5 to 3.0]

8. Primary Outcome: Tmax for Benzyl Alcohol
Description: The time after administration of Natroba (spinosad) Topical Suspension, 0.9% when the maximum plasma concentration is reached for benzyl alcohol.
Time Frame: as for outcome 1
Population: Per Protocol
Measure: Median (Full Range); unit: hours
Arm/Group | Natroba
Number analyzed (Participants) | 26
hours | 0.5 (0.3071) [0.5 to 3.0]

9. Primary Outcome: AUC (0-12) for Benzyl Alcohol
Description: Area under the plasma concentration versus time curve (AUC) of benzyl alcohol in Natroba (spinosad) Topical Suspension, 0.9%.
Time Frame: as for outcome 1
Population: Since the only benzyl alcohol concentrations above Limit of Quantitation (LOQ) (1.0 μg/mL) were for 1 sample each for 4 subjects and 2 non-consecutive samples for 2 subjects, AUC (0-12) was not summarized.
Measure: Number; unit: μg*hr/mL
Arm/Group | Natroba
Number analyzed (Participants) | 26
μg*hr/mL | NA — Since the only benzyl alcohol concentrations above LOQ (1.0 μg/mL) were for 1 sample each for 4 subjects and 2 non-consecutive samples for 2 subjects, AUC 0-12 was not summarized.

ADVERSE EVENTS:
Time Frame: Throughout the study.
Description: All Adverse Events (AEs)occurring during the study were recorded at 0 (pretreatment), 0.5, 1, 3, 6, and 12 hours post-treatment by age group and all subjects. Verbatim descriptions of AEs were assigned to system organ classes and preferred terms using the Medical Dictionary for Regulatory Activities (MedDRA) (v14.0).
Arm/Group | Natroba
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 9/26
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natroba (N=26)
Pyrexia (General disorders) | 7 (13)
Application Site Pruritus (General disorders) | 3 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (13)
Erythema (Skin and subcutaneous tissue disorders) | 1 (13)

LIMITATIONS AND CAVEATS:
It is suspected for Subject 02-202, at 0.5 hours, the sample to determine the spinosyn A and spinosyn D concentrations were possibly contaminated with Natroba.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No